CLINICAL TRIAL: NCT02983929
Title: Impact of Elevated Body Mass Index on Short-term Follow-up Indicators for Total Knee Arthroplasty : a Retrospective Study
Brief Title: Short-Term Follow-up Indicator for Total Knee Arthroplasty and Body Mass Index
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Durécu Lavoisier (Other)
Responsible Party: Principal Investigator, Timothée Gillot, Physical therapist, Msc., Centre Hospitalier Durécu Lavoisier
Other Study IDs: MK1
Record Dates: First submitted 2016-11-29; First posted 2016-12-06 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Total Knee Arthroplasty; Body Mass Index; Rehabilitation

STUDY DESIGN:
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BMI <30 kg.m-2: Patients with a BMI inferior to the obesity limit defined by the World Health Organization.
  Interventions: Procedure: Rehabilitation after total knee arthroplasty
- BMI >30 kg.m-2: Patients with a BMI superior to the obesity limit defined by the World Health Organization.
  Interventions: Procedure: Rehabilitation after total knee arthroplasty

INTERVENTIONS:
Procedure: Rehabilitation after total knee arthroplasty — All the included patients followed a rehabilitation program in the Polyvalent Geriatric Rehabilitation Clinic after total knee arthroplasty.

SUMMARY:
The main purpose of this study is to determine the influence of obesity on the short term follow-up indicators of a polyvalent geriatric rehabilitation clinic after total knee arthroplasty. It is a retrospective, comparative study

The secondary purposes are to explore the links between length of stay and short-term follow-up indicators of a polyvalent geriatric rehabilitation clinic after total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted after total knee arthroplasty in Polyvalent Geriatric Rehabilitation Clinic during the january 2007/October 2016 period

Exclusion Criteria:

* Uncompleted case file or case file anterior to 2007 ;
* Inter-current orthopedic complication ;
* Evolutive or inter-current pathology written in the case-file (neurologic affection, etc...).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men and Women admitted after total knee arthroplasty in Polyvalent Geriatric Rehabilitation Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2007-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 2 Month
Range Of Motion of the Knee | 2 Month
  The investigators will report the initial, final flexion and extension and calculate the total gain of flexion and extension of the knee for each participant.
Age | 2 Month
Mansat Score | 2 Month
  This score is a composite score recommended by the French Authority of Health.

SECONDARY OUTCOMES:
Length of stay | 2 month
  The investigators will report the length of stay in the rehabilitation clinic for each participant.